CLINICAL TRIAL: NCT06876610
Title: Application of CfDNA Methylation Detection in Auxiliary Diagnosis of Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Geneplus-Beijing Co. Ltd. (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 25/071-5017
Record Dates: First submitted 2025-03-07; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Screening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Cancer Arm: Participants with breast cancer from which a tumor tissue will be collected. Participants with new diagnosis of breast cancer from which a blood sample will be collected.
- Benign Diseases Arm: Participants with breast benign diseases from which a tissue will be collected. Participants with breast benign diseases from which a blood sample will be collected.

SUMMARY:
The purpose of this study is to construct an auxiliary diagnostic model for breast cancer by methylation markers. The study will collect blood and tissue samples from participants with breast cancer and benign disease for whole-genome methylation sequencing. It will screen methylation markers and develop a methylation auxiliary diagnosis model to distinguish between breast cancer and non-cancer.

ELIGIBILITY:
Inclusion Criteria for All the Participants:

* With confirmed pathological diagnosis and molecular subtyping results
* Ability to provide a written informed consent

Exclusion Criteria for Cancer Arm Participants:

* Patients with a history of or currently suffering from other malignancies
* Pregnant or planning to become pregnant female patients
* Patients who have received cancer treatment, including surgery, chemotherapy, radiotherapy, targeted therapy, and immunotherapy, before blood draw
* Patients with a history of blood transfusion within the past month
* Patients with a known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
* Patients with persistent fever or undergoing anti-inflammatory treatment within 14 days before blood draw
* Any other conditions that the researcher deems may make the patient unsuitable for inclusion in the study or may interfere with the completion of the study
* Patients in poor physical condition who are not suitable for blood draw
* Patients who cannot provide informed consent or refuse blood draw

Exclusion Criteria for Benign Diseases Arm Participants:

* History of malignancies
* Current malignancies or precancerous lesions

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from medical centers and assigned into two arms, including participants with new diagnosis of breast cancer and benign diseases.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Establish DNA methylation profiles of two populations by collecting tissues and peripheral blood related to benign and malignant breast nodules. | 12 months
Based on DNA methylation profiles, systematically evaluate the signal, noise, and complementarity of methylation biomarkers and ultimately form a set of diagnostic biomarker combinations for breast malignant nodules. | 12 months
Further develop a methylation assisted diagnostic model that can effectively distinguish between benign and malignant breast nodules. | 12 months

SECONDARY OUTCOMES:
Evaluate the contribution and performance of methylation assisted diagnostic models by integrating imaging and methylation assisted diagnostic model results, and clarify the specificity and sensitivity of integrated model diagnosis. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China